CLINICAL TRIAL: NCT05919316
Title: The Efficacy Of Rhinophototherapy Compared To Intranasal Corticosteroids On The Nasal Mucosa Of Allergic Rhinitis Patients
Brief Title: The Efficacy Of Rhinophototherapy Compared To Intranasal Corticosteroids On The Nasal Mucosa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GGPM-2022-028
Record Dates: First submitted 2023-06-16; First posted 2023-06-26 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Mometasone Furoate

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhinophototherapy (Experimental): Intranasal Rhinophototherapy is an electronic allergic rhinitis treatment device (brand Bionette) also a medical device that producing low level narrow band red light at a wavelength of 630nm. It is a Class B medical device (registration of Malaysia number GB67793908818). It is powered by two alkaline button batteries with a dimension of 52mm x 40mm and weighing less than 20g . Light is produced via nasal prongs which are to be inserted into both nostrils. Plastic nasal cannula are available and can be replaced to ensure sterility and prevent transmission of infection.
  Interventions: Device: Rhinophototherapy
- Intranasal Corticosteroids (Active Comparator): Mometasone furoate will be available in the form of Nasonex Nasal Spray. It has a dose of 50 mcg/dose mometasone furoate per spray, registration no: MAL20001010AZ, distributed by: Merck Sharp & Dohme (Malaysia) Sdn. Bhd.
  Interventions: Drug: Nasonex Nasal Spray

INTERVENTIONS:
Device: Rhinophototherapy — Intranasal rhinophotometer to be used at home for 4.5 minutes three times daily for 14 days
  Other Names: Intranasal rhinophototherapy Bionette
  Arms: Rhinophototherapy
Drug: Nasonex Nasal Spray — 50mcg/dose, 2 sprays each nostril (morning or evening) once daily for 14 days
  Other Names: Mometasone furoate nasal spray
  Arms: Intranasal Corticosteroids

SUMMARY:
The aim of this study to compare the efficacy of Rhinophototherapy to Intranasal Corticosteroids on the the nasal mucosa of allergic rhinitis patients. The main question to answer is: Does intranasal phototherapy reduce inflammation in the tissue biopsy of the inferior turbinate mucosa compared to intranasal steroids?

The hypothesis for this study is Intranasal phototherapy will reduce mucosal inflammation without mucosal damage and is comparable to intranasal steroids in allergic rhinitis patients

DETAILED DESCRIPTION:
There are several specific objectives for this study:

1. To subjectively and objectively compare the efficacy of intranasal phototherapy and intranasal corticosteroids in treating allergic rhinitis via assessment of rhinomanometry, peak nasal inspiratory flow (PNIF) and visual analogue scale(VAS) score.
2. To determine mucosal inflammatory cells changes (eosinophils, neutrophils, mast cells) between patients treated with intranasal rhinophototherapy and intranasal corticosteroids.
3. To determine mucosal damage (fibrosis, mucosal ulceration , squamous metaplasia) between patients treated with intranasal rhinophototherapy and intranasal corticosteroids.

Patients who meet the criteria to join the study will be randomized in a single-blinded manner(investigator). Patients will be given information about the study and consent form, patients will be randomized to 2 treatment group (rhinophototherapy and Nasonex nasal spray). Patients will be evaluated before and after treatment in two weeks time.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years and above
* Newly diagnosed allergic rhinitis
* Allergic rhinitis is confirmed via positive skin prick test or serum Immunoglobulin E

Exclusion Criteria:

* Anaphylaxis /poorly controlled bronchial asthma
* Refused nasal biopsy
* Usage of intranasal corticosteroids and/or antihistamine sprays for the past 1 month
* Consumption of oral leukotriene receptor antagonist or oral steroids for the past 1 month
* Concomitant nasal pathology (malignancy, chronic rhinosinusitis with nasal polyposis, severe deviated nasal septum)
* Bleeding disorder or on anticoagulant/antiplatelet therapy
* Recent URTI/Covid-19 within past 14 days
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Symptoms Score of Allergic Rhinitis at week 2 | Baseline and Week 2
  The Visual Analogue Score (VAS) is a validated, self-reported instrument assessing average scoring of overall allergic rhinitis symptoms and details of allergic symptoms (runny nose, sneezing, nasal blockage, nasal itchiness) in the last 14 days period from treatment date. Possible score range from 0 (no symptoms) to 100 (worst possible symptoms). Maximum number of change from baseline indicate improvement of symptoms.
  Change= (Baseline score - Week 2 score)
Peak nasal inspiratory flow meter (PNIF) | Baseline and Week 2
  PNIF is an easy to use object which measures airflow through the nose during maximal inspiration. Air flow is measured via a variable diameter in litre/minute. Inertia of inspiratory air will move the marker to indicate the maximum flow achieved. The best of 3 attempts of inspiration will be taken. The maximum value indicates better result of inspiration.
Total nasal resistance by Rhinomanometry | Baseline and Week 2
  Rhinomanometry provides a functional measure of pressure/flow during a breathing cycle. It is to be performed at week 0, prior to commencement of nasal spray and week 2 of treatment for comparisons. Normal values for total nasal resistance is below 0.2 and to 0.3 Pa cm3/s. Worst case will be higher than 0.3 Pa cm3/s indicate nasal obstruction.
  Change= (Baseline score - Week 2 score)
Determination of mucosal inflammatory cells changes (eosinophils, neutrophils, mast cells) between patients treated with intranasal rhinophototherapy and intranasal corticosteroids. | Week 2
  Nasal mucosa biopsy will be performed after 2 weeks of usage of intranasal phototherapy/corticosteroids under local anesthesia. Biopsy samples will be kept in glass bottles filled with paraformaldehyde. It will be labelled, packaged with a biohazard wrap and be transported within an hour to the histopathology lab.
  Quantification of eosinophil, neutrophil and mast cell numbers in inferior turbinate tissue biopsy will be performed by counting numbers of stained cells. Results are expressed as the number of cells per one hpf of tissue.
Determination of mucosal damage (fibrosis, mucosal ulceration , squamous metaplasia) between patients treated with intranasal rhinophototherapy and intranasal corticosteroids. | Week 2
  Nasal mucosa biopsy will be performed after 2 weeks of usage of intranasal phototherapy/corticosteroids under local anesthesia. Biopsy samples will be kept in glass bottles filled with paraformaldehyde. It will be labelled, packaged with a biohazard wrap and be transported within an hour to the histopathology lab.
  Tissue will be assessed histologically based on a modified grading system.
  Mucosal damage:
  * mucosal ulceration (absent or present)
  * squamous metaplasia (absent or present)
  * Presence of fibrosis (absent or present)

CONTACTS AND LOCATIONS:
Overall Officials: Hardip Singh Gendeh, Principal Investigator — Otorhinolaryngology Department, Head and Neck Surgery, Faculty of Medicine, UKM Medical Centre
Locations (1):
- Otorhinolaryngology Department, Head and Neck Surgery, Faculty of Medicine, UKM Medical Centre, Jalan Yaacob Latif, Bandar Tun Razak, Cheras, Kuala Lumpur, Cheras, Malaysia

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication plan to be shared to researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research.

REFERENCES:
- [Derived] Ramasamy K, Gendeh HS, Wan Hamizan AK, Md Pauzi SH, Zahedi FD, Megat Ismail NF, Alfian N, Abdul Razak NN, Chinna K, Husain S. Histological Impact of Rhinophototherapy Compared to Intranasal Corticosteroids on Inflammatory Cells and Nasal Mucosa in Allergic Rhinitis. Ann Otol Rhinol Laryngol. 2026 Jan 7:34894251401132. doi: 10.1177/00034894251401132. Online ahead of print. PMID 41501617